CLINICAL TRIAL: NCT01830335
Title: The Influence of Cerebral Blood Flow and Alkalosis on Neuromuscular Function During Environmental Stress
Brief Title: Cerebral Blood Flow and PETCO2 on Neuromuscular Function During Environmental Stress
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Stephen Cheung, Professor, Brock University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-167
Record Dates: First submitted 2013-03-20; First posted 2013-04-12 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Healthy Males; Neuromuscular Function
MeSH Terms: interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental): Indomethacin 1.2 mg kg 1 dose
  Interventions: Drug: Indomethacin
- Placebo (Placebo Comparator): flour capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Indomethacin
  Arms: Drug
Drug: Placebo
  Arms: Placebo

SUMMARY:
Environmental stress, such as low oxygen availability (hypoxia), has been associated with impaired neuromuscular performance; however, the mechanisms associated with these performance decrements remain unclear. While the majority of research suggests that the observed fatigue is related to the central nervous system, the influence of changes in cerebral blood flow (CBF) and associated changes in cerebral pH (partial pressure of carbon dioxide; PCO2) remains unexamined. In response to hypoxic stress, humans hyperventilate to maintain oxygen consumption, resulting in a hypocapnia mediated decrease in CBF and cerebral alkalosis (decreased PCO2). Previous research suggests that hyperventilation induces changes in neural excitability and synaptic transmission; however, it remains unclear if these changes are related to hypocapnia mediated decrease in CBF or cerebral alkalosis or both.

The purpose of the proposed research program is to examine the influence of changes in CBF and cerebral alkalosis on neuromuscular function during environmental stress. The research program will consist of 2 separate projects, summarized below in a table outlining the proposed protocols and resultant physiological manipulations. During each manipulation, neuromuscular function will be evaluated and compared to baseline (normoxic) conditions using a repeated measures design.

The research program will consist of 2 separate projects. Project 1 will examine the changes in CBF and alkalosis by using (a) indomethacin (decrease CBF; no change PCO2) and (b) hypocapnia (decrease CBF; decrease PCO2). Using a similar experimental design, Project 2 will examine the change in CBF and alkalosis during hypoxia by using (a) poikilocapnic hypoxia (decrease PO2; decrease CBF; decrease PCO2), (b) isocapnic hypoxia (decrease PO2; no change CBF; no change PCO2) and (c) isocapnic hypoxia + indomethacin (decrease PO2; decrease CBF; no change PCO2). During each manipulation, neuromuscular function will be evaluated and compared to baseline (normoxic) conditions using a repeated measures design.

Therefore, Project 1 will examine the separate and combined effect of changes in CBF and cerebral alkalosis on neuromuscular function independent of environmental manipulations. Subsequently, Project 2 will examine neuromuscular function during hypoxia while controlling CBF and cerebral alkalosis. It is hypothesized that changes in PCO2 and therefore, changes in cerebral alkalosis will contribute to neuromuscular fatigue independent of changes in CBF and oxygen availability.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 25 yrs old; healthy males

Exclusion Criteria:

* diagnosed medical condition; NSAID allergy; smoker; high altitude exposure; implants

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Resting motor threshold | Change from baseline 90-minutes
  Motor evoked potentials are recorded from muscles following transcranial magnetic stimulation of motor cortex. The resting motor threshold is defined as the minimum stimulation intensity required to elicit a motor evoked potential. Resting motor threshold will be quantified in millivolts.
H-Reflex Amplitude | Change from baseline 90-minutes
  The H-Reflex is an indirect measure of motor neuron excitability. Initially, a maximal M-wave (M-max) will be elicited by stimulating (1 ms in duration; 15 s between stimuli) the median nerve incrementally (2 V increments) until the largest waveform is observed. The peak-to-peak amplitude of this waveform is considered M-max. Using similar procedures as above, a sub-maximal M-wave of 5% M-max will be elicited and the amplitude of the resultant H-reflex (a small waveform observed following the submaximal M-wave) will be calculated. The amplitude of the H-reflex will be quantified in milllivolts.
Maximal Voluntary Contraction | Change from baseline 90-minutes
  During maximal voluntary contraction (MVC) testing, the participants' right arm will be secured in a custom made device used to isolate forearm flexion and to measure force production by the flexor carpi radialis muscle. Participants will be asked to produce a 5-second MVC and will be verbally encouraged to maintain maximal force production throughout the duration of the contraction. MVC will be quantified as the maximum force production in newton meters.
H-reflex latency | Change from baseline 90-minutes
  The H-Reflex is an indirect measure of motor neuron excitability. Initially, a maximal M-wave (M-max) will be elicited by stimulating (1 ms in duration; 15 s between stimuli) the median nerve incrementally (2 V increments) until the largest waveform is observed. The peak-to-peak amplitude of this waveform is considered M-max. Using similar procedures as above, a sub-maximal M-wave of 5% M-max will be elicited and the amplitude of the resultant H-reflex (a small waveform observed following the submaximal M-wave) will be calculated. The onset latency of the H-reflex will be quantified in milliseconds.
Voluntary Activation | Change from baseline 90-minutes
  The level of neural drive to muscle during contraction is termed voluntary activation and will be estimated by interpolation of a single supramaximal motor evoked potential during the 5-second MVC contraction. If extra force is evoked by the 'superimposed' stimulus then either the stimulated axons were not all recruited voluntarily or they were discharging at sub-tetanic rates. Therefore, voluntary activation will be quantified as the amplitude of maximal voluntary force production, relative to the amplitude of the supramaximal MEP.

SECONDARY OUTCOMES:
Middle Cerebral Artery Blood Flow Velocity | Change from baseline 90-minutes
  Middle cerebral artery (MCA) blood flow velocity will be measured non-invasively by a 2-MHz transcranial Doppler (TCD) ultrasound probe, attached bilaterally to a comfortable headband and secured anterior to the zygomatic arch, rostral of the pinna. Doppler probes will be paced over the temporal windows (near the ear) and will remain in place throughout the duration of the experimental protocol. MCA velocity will be quantified in cm/s.
Brachial Artery Blood flow | Change from baseline 90-minutes
  Brachial artery blood flow will be measured non-invasively using a high-resolution ultrasound machine. Participants will lie supine with their forearm extended in a comfortable position. Blood flow measurements will be taken in the top 1/3 of the upper arm over the duration of 10 cardiac cycles (approximately 60 seconds). Blood flow will be quantified in L/min.
Internal Carotid Artery Blood Flow | Change from baseline 90-minutes
  Internal carotid artery (ICA) blood flow will be measured non-invasively using a high-resolution ultrasound machine. Participants will lie supine with a slight extension of the neck and at 45° of lateral flexion away from the side being scanned. ICA measurements will be taken 1 cm superior to the common carotid bifurcation over the duration of 10 cardiac cycles (approximately 60 seconds). Blood flow will be quantified in L/min.
Blood pressure | Change from baseline 90-minutes
  Beat by beat blood pressure will be calculated from the blood pressure waveform using finger photoplethysmography (Nexfin, bmeye), with a finger cuff placed directly over the middle finger on the left hand. Blood pressure will be quantified in mmHg.
Pulse oximetry | Change from baseline 90-minutes
  A pulse oximetry probe will be placed over a finger to provide a continuous, non-invasive measurement of the blood oxygen saturation to confirm that the end-tidal forcing system is controlling oxygen delivery at the desired levels during each experiment. Oxygen saturation will be quantified as a percentage.
Heart Rate | Change from baseline 90-minutes
  Heart rate will be measured by electrocardiogram. Heart rate will be quantified in beats per minute.
End-Tidal Gas Concentrations | Change from baseline 90-minutes
  The end-tidal concentrations of oxygen and carbon dioxide will be measured and reported in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cheung, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada